CLINICAL TRIAL: NCT04518319
Title: Clinical Comprehensive Intervention on Cognitive Impairment of Schizophrenia Patients With Metabolic Syndrome
Brief Title: Clinical Intervention on Cognitive Impairment of Schizophrenia With Metabolic Syndrome
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: The COVID-19 affects the recruitment of patients.
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, Yan CHEN, PI, Shanghai Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20200815SMHC-sk-YChen
Record Dates: First submitted 2020-08-13; First posted 2020-08-19 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Docosahexaenoic Acids; Transcranial Direct Current Stimulation; Olanzapine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- omega-3 polyunsaturated fatty acids (Experimental): Patients randomized to the omega-3 polyunsaturated fatty acids will receive treatment with 1200mg per day plus on-going olanzapine.
  Interventions: Drug: Omega-3 polyunsaturated fatty acids
- Xbox aerobic exercise (Experimental): Patients randomized to the Xbox aerobic exercise will do Xbox aerobic exercise 30min per day plus on-going olanzapine.
  Interventions: Behavioral: Xbox aerobic exercise
- transcranial direct current stimulation (Experimental): Patients randomized to the transcranial direct current stimulation will be applied for transcranial direct current stimulation 5 session/week at 2mA, 20min plus on-going olanzapine. The anodal electrode will be placed over the left dorsolateral prefrontal cortex.
  Interventions: Device: transcranial direct current stimulation,tDCS
- olanzapine (Experimental): Patients randomized to the olanzapine will receive conventional treatment-olanzapine.
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Omega-3 polyunsaturated fatty acids — Omega-3 polyunsaturated fatty acids will be taken 1200mg per day plus on olanzapine.
  Arms: omega-3 polyunsaturated fatty acids
Behavioral: Xbox aerobic exercise — Patients will do Xbox aerobic exercise 30min per day plus on olanzapine.
  Arms: Xbox aerobic exercise
Device: transcranial direct current stimulation,tDCS — Patients will receive tDCS at 2mA, 20 min for 5 session per week plus on olanzapine.
  Arms: transcranial direct current stimulation
Drug: Olanzapine — Patients will take only olanzapine pills.
  Arms: olanzapine

SUMMARY:
This is a single-center, randomized, parallel-control study conducted in schizophrenic inpatients with metabolic syndrome who have been conducted with olanzapine. The purpose of this study is to evaluate the efficacy and safety of omega-3 polyunsaturated fatty acids, Xbox aerobic exercise and transcranial direct current stimulation( tDCS). Following a screening period, subjects who meet the entry criteria will be randomized to treated with omega-3 polyunsaturated fatty acids1.2mg per day, Xbox aerobic exercise 30min per day and tDCS at 2mA, 20 min(5 session/week) for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Meets the Diagnostic and Statistical Manual of Mental Disorder,Fifth Edition(DSM-V) criteria for Schizophrenia.
2. Patients have got standard treatment of olanzapine monotherapy for more than 6 months, PANSS baseline ≤ 60.
3. Meets the ATP-III criteria for metabolic syndrome.
4. Male or female subjects aged 18-60 years, education level of junior high school for above.
5. The patient fully understand and signed the informed consent form.

Exclusion Criteria:

1. Serious and instable body disease such as cerebrovascular disease, liver and kidney disease, disease of internal secretion (abnormal thyroid function), blood disease; any history of seizures or other organic brain diseases.
2. Pregnant or lactating women and women of childbearing potential throughout the study period; patients who have plans to move to other places within the year.
3. History of diabetes, hyperlipidemia and other metabolic abnormalities.
4. Due to other reasons, the researchers considered it unsuitable to participate in this clinical trial.

   -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Explore the treatment of cognitive impairment in schizophrenia patients with metabolic syndrome | from baseline to 3 months after treatment
  Change in the the MATRICS consensus cognitive battery between randomization

SECONDARY OUTCOMES:
change in the Schizophrenia Quality of Life Scale(SQLS) | assessed from baseline to 3 months after treatment
  The aim is to explore what kind of intervention will improve the quality of life as measured with the Schizophrenia Quality of Life Scale(SQLS). The scores between 1-100. The lower scores means a better outcome.
change in the scale of social function in psychosis inpatients | assessed from baseline to 3 months after treatment
  The aim is to explore what kind of intervention will improve the patients' social function as measured with the scale of social function in psychosis inpatients(SSPI).<18 points means severe defects, 18-28 points means moderate defects, 29-38 means mild defects. The higher scores means a better outcome.
metabolic indicators | assessed from baseline to week 24
  Height(kilograms) and weight(meters) will be measured to evaluate the patients' BMI(kg/m2) at baseline, week4,12,16(1months after treatment ) and 24(3 months after treatment).
biological index | assessed from baseline to week 24
  CRP(mg/dl) will be tested to determine whether the interventions measures will affect the inflammatory biomarkers.
biological index | assessed from baseline to week 24
  C3（g/l）will be tested to determine whether the interventions measures will affect the inflammatory biomarkers
biological index | assessed from baseline to week 24
  IL-6(U/L) will be tested to determine whether the interventions measures will affect the inflammatory biomarkers.
biological index | assessed from baseline to week 24
  brain-derived neurotrophic factor( BDNF) will be tested to determine whether the interventions measures will affect the BDNF.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Chen, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China